CLINICAL TRIAL: NCT00413166
Title: Treatment of Acute Promyelocytic Leukemia (APL) With All-Trans Retinoic Acid, and Arsenic +/- Idarubicin
Brief Title: All-trans Retinoic Acid, and Arsenic +/- Idarubicin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0706; NCI-2012-01395 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-12-15; First posted 2006-12-19 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Acute Promyelocytic Leukemia; APL; ATRA; All-Trans Retinoic Acid; Arsenic Trioxide; Theophylline; Gemtuzumab
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Tretinoin; Arsenic Trioxide; Idarubicin; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Induction ATRA + ATO + Idarubicin (Experimental): All-Trans Retinoic Acid (ATRA) + Arsenic Trioxide (ATO)
  ATRA 45 mg/m2 daily by mouth beginning day 1; ATO 0.15 mg/kg by vein daily beginning on day 1; Idarubicin 12 mg/m2 x 1 dose; Methylprednisolone 50 mg daily for 5 days starting on day 1.
  Interventions: Drug: All-Trans Retinoic Acid (ATRA); Drug: Arsenic Trioxide (ATO); Drug: Idarubicin
- Maintenance (Experimental): All-Trans Retinoic Acid (ATRA) + Arsenic Trioxide (ATO)
  ATO 0.15 mg/kg by vein over 2 hours Monday-Friday for 4 weeks, then a 4-week break. ATRA 45 mg/m2 by mouth every day for 2 weeks, followed by 2 additional weeks of no study drug. Continue ATRA until treatment with ATO complete.
  Interventions: Drug: All-Trans Retinoic Acid (ATRA); Drug: Arsenic Trioxide (ATO); Drug: Idarubicin
- Induction ATRA + ATO + GO (Experimental): All-Trans Retinoic Acid (ATRA) + Arsenic Trioxide (ATO) + Gemtuzumab Ozogamicin (GO)
  ATRA 45 mg/m2 daily po (in 2 divided doses) beginning day 1; ATO 0.15 mg/kg IV daily beginning on day 1; GO 9 mg/m2 on day 1 Methylprednisolone 50 mg daily for 5 days followed by rapid taper starting on day 1.
  Theophylline 100mg p.o. bid days 1-3, 200 mg p.o. bid days 4-6, and 300 mg p.o. bid thereafter during periods when patient is receiving ATRA or ATO. Theophylline administration continues until therapy with ATO and ATRA is completed.
  Interventions: Drug: All-Trans Retinoic Acid (ATRA); Drug: Arsenic Trioxide (ATO); Drug: Idarubicin; Drug: Gemtuzumab Ozogamicin

INTERVENTIONS:
Drug: All-Trans Retinoic Acid (ATRA) — Induction: 45 mg/m2 daily by mouth in 2 divided doses beginning day 1
Drug: Arsenic Trioxide (ATO) — Induction: 0.15 mg/kg daily IV beginning day 1
Drug: Idarubicin — 1. 12 mg/m2 one dose only (may be given on day 1 to 5 of induction)
  2. If either ATRA or ATO are discontinued due to toxicity, idarubicin 12 mg/m2 x 2 doses will be administered once every 4 to 5 weeks (depending on the recovery of counts) until 28 weeks has elapsed from the Complete Recovery date.
  Other Names: Idamycin
Drug: Gemtuzumab Ozogamicin — Induction: 9 mg/m2 on day 1 of induction
  Arms: Induction ATRA + ATO + GO

SUMMARY:
The goal of this clinical research study is to learn if the combination of arsenic trioxide (ATO) with ATRA and possibly idarubicin is effective in treating patients with newly-diagnosed APL.

DETAILED DESCRIPTION:
All-trans retinoic acid (ATRA) and ATO are designed to cause the APL cells to mature and function normally. Idarubicin is designed to cause breaks in both strands of DNA (the genetic material of cells).

If you are found to be eligible to take part in this study, you will begin induction. During induction, you will receive ATRA, by mouth starting on Day 1. You will also receive ATO through a needle in your vein over 2 hours starting on Day 1. You will continue receiving the drugs every day until your bone marrow no longer shows APL cells.

If you had a high white blood cell count at screening, you will receive idarubicin through a needle in your vein over about 30 minutes one dose only on any day of Day 1 through 5.

During induction, blood (about 1-3 tablespoons) will be drawn every day during Week 1, and then 2 times a week after that. This blood will be drawn for routine tests.

During induction (about 21-28 days after beginning treatment), you will have a bone marrow aspirate to check the status of the disease. This may be performed more often if the doctor thinks it is needed.

If you achieve a complete remission during the induction phase, you will continue to the maintenance phase. During the maintenance phase, you will receive ATO by vein over 2 hours Monday-Friday for 4 weeks. After the 4 weeks of receiving the study drug, you will have a 4-week period "off" (when no study drug is given). ATRA is given by mouth every day for 2 weeks. This 2 weeks is followed by 2 additional weeks when no study drug will be given. You will continue to take ATRA until treatment with ATO is complete.

During maintenance, blood (about 1-3 tablespoons) will be drawn before every 4-week cycle of ATO, and then every week for routine tests. You will also have an ECG before every 4 week cycle when you take ATO.

If you do not achieve a complete remission during induction you will be taken off study.

If at any point during the study your white blood cell count rises above 10,000, you will receive idarubicin by vein over 30 minutes.

You will remain in the hospital for about the first 7 days of induction. After that, you must remain in Houston for the next 3-4 weeks. Once in the maintenance phase, you may be treated at home, but must return to M. D. Anderson for study visits.

After maintenance is complete, you will have follow-up visits for an additional 2 years. If at any time during the active study or follow-up the disease gets worse or intolerable side effects occur, you will be taken off the study.

If you had a low or high white blood cell count when you joined the study, you will have follow-up visits every 3 months for 2 years. At these visits, blood (about 1 tablespoon) will be drawn for routine tests and you will have a bone marrow aspirate.

This is an investigational study. Idarubicin, ATRA and ATO are FDA approved and commercially available. However, their use in this study and in this combination is considered investigational. Its use in APL patients is investigational. Up to 80 patients will take part in this multicenter study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of APL based on the presence of the PML-RAR alpha fusion gene by cytogenetics, PCR, or POD test.
2. Provision of written informed consent.
3. Patients in whom therapy for APL was initiated on an emergent basis are eligible

Exclusion Criteria:

1. First trimester of pregnancy (ATRA is teratogenic)
2. Corrected QT (QTC) interval must not be greater than 480 milliseconds.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 5, 2006 to April 3, 2012. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Pfizer withdrew gemtuzumab ozogamycin (GO) from market based Food & Drug Administration recommendation. As such, protocol modified to Idarubicin Day 1 of induction in high-risk participants & in low risk participants with rising white blood count (WBC), Idarubicin administered to low-risk patients in whom WBC >10,000 after initiation of ATRA + ATO.
Groups:
- ATRA + ATO: Low Risk (WBC<10,000): All-Trans Retinoic Acid (ATRA) + Arsenic Trioxide (ATO): Oral ATRA 45 mg/m2 daily beginning day 1; ATO 0.15 mg/kg by vein (IV) daily beginning day 1; Idarubicin 12 mg/m2 x 1 dose; Methylprednisolone 50 mg daily for 5 days. Methylprednisolone 500 mg daily for 5 days followed by rapid taper starting on day 1
  Idarubicin: 1) 12 mg/m2 one dose only (day 1 to 5 of induction) as needed for WBC>10,000. 2) If ATRA or ATO discontinued due to toxicity, idarubicin 12 mg/m2 x 2 doses administered once every 4- 5 weeks until 28 weeks elapsed from Complete Recovery date.
  Post CR
  1.) ATO 0.15 mg/kg IV for 5 of every 7 days on each of weeks 1-4 (course 2), 9-12 (course 3), 17-20 (course 4), and 25-28 (course 5) (thus 4 courses). 2.) Oral ATRA 45 mg/m2 daily on a "2-weeks on -2-weeks off" basis until therapy with ATO completed.
- ATRA+ATO+IDA: High Risk (WBC >10,000): Oral ATRA 45 mg/m2 daily beginning day 1; ATO 0.15 mg/kg IV daily beginning day 1; Idarubicin (IDA) 12 mg/m2 x 1 dose; Methylprednisolone 50 mg daily for 5 days.
  ATRA Induction: 45 mg/m2 daily by mouth in 2 divided doses beginning day 1; and ATO: Induction: 0.15 mg/kg daily IV beginning day 1.
  Idarubicin: 1) 12 mg/m2 one dose only (day 1 to 5 of induction) 2) If ATRA or ATO discontinued due to toxicity, idarubicin 12 mg/m2 x 2 doses administered once every 4- 5 weeks until 28 weeks elapsed from Complete Recovery date.
- ATO+ATRA+GO: ATRA 45 mg/m2 daily po (in 2 divided doses) beginning day 1 ATO 0.15 mg/kg IV daily beginning on day 1 Methylprednisolone 50 mg daily for 5 days followed by rapid taper starting on day 1 GO 9 mg/m2 on day 1 of induction Theophylline 100mg p.o. bid days 1-3, 200 mg p.o. bid days 4-6, and 300 mg p.o. bid thereafter during periods when patient is receiving ATRA or ATO. Theophylline administration continues until therapy with ATO and ATRA is completed.
  Post-CR treatment ATO 0.15 mg/kg IV over 2 hours Monday-Friday for 4 weeks, then 4-week break. Oral ATRA 45 mg/m2 every day for 2 weeks, followed by 2 additional weeks of no study drug. Continue ATRA until treatment with ATO complete.
Period: Overall Study
Arm/Group | ATRA + ATO: Low Risk (WBC<10,000) | ATRA+ATO+IDA: High Risk (WBC >10,000) | ATO+ATRA+GO
Started | 57 | 5 | 16
Completed | 57 | 5 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ATO+ATRA+GO: Induction ATRA 45 mg/m2 daily po (in 2 divided doses) beginning day 1 ATO 0.15 mg/kg IV daily beginning on day 1 Methylprednisolone 50 mg daily for 5 days followed by rapid taper starting on day 1 GO 9 mg/m2 on day 1 of induction Theophylline 100mg p.o. bid days 1-3, 200 mg p.o. bid days 4-6, and 300 mg p.o. bid thereafter during periods when patient is receiving ATRA or ATO. Theophylline administration continues until therapy with ATO and ATRA is completed.
  Post-CR treatment ATO 0.15 mg/kg IV over 2 hours Monday-Friday for 4 weeks, then 4-week break. Oral ATRA 45 mg/m2 every day for 2 weeks, followed by 2 additional weeks of no study drug. Continue ATRA until treatment with ATO complete.
- Total: Total of all reporting groups
Arm/Group | ATRA + ATO: Low Risk (WBC<10,000) | ATRA+ATO+IDA: High Risk (WBC >10,000) | ATO+ATRA+GO | Total
Number analyzed (Participants) | 57 | 5 | 16 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 46 | 5 | 15 | 66
  >=65 years | 10 | 0 | 1 | 11
Age, Continuous [Median (Full Range); unit: years] | 49 [16 to 84] | 38 [28 to 63] | 44 [19 to 75] | 47 [16 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 2 | 12 | 47
  Male | 24 | 3 | 4 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 1 | 4 | 11
  White | 46 | 2 | 12 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 57 | 5 | 16 | 78

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate
Description: Response defined as CR (marrow with <5% blasts and no abnormal promyelocytes together with neutrophil count >1000 and platelet count >100,000) and toxicity as Acute promyelocytic leukemia (APL) differentiation syndrome, arrhythmia, peripheral neuropathy.
  Bone marrow aspirate performed to check the status of the disease.
Time Frame: 1 month, up to day 85 of treatment
Population: Of the 57 participants treated on the ATRA + ATO: Low Risk treatment arm, 56 participants were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | ATRA + ATO: Low Risk (WBC<10,000) | ATRA+ATO+IDA: High Risk (WBC >10,000) | ATO+ATRA+GO
Number analyzed (Participants) | 56 | 5 | 16
Participants | 55 | 5 | 15

ADVERSE EVENTS:
Time Frame: Up to 7 years
Arm/Group | ATRA + ATO: Low Risk (WBC<10,000) | ATRA+ATO+IDA: High Risk (WBC >10,000) | ATO+ATRA+GO
All-Cause Mortality (participants affected / at risk) | 1/57 | 0/5 | 1/16
Serious Adverse Events (participants affected / at risk) | 22/57 | 4/5 | 4/16
Other Adverse Events (participants affected / at risk) | 5/57 | 0/5 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATRA + ATO: Low Risk (WBC<10,000) (N=57) | ATRA+ATO+IDA: High Risk (WBC >10,000) (N=5) | ATO+ATRA+GO (N=16)
Appendectomy (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Troponin I (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed level of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated Transaminases (Metabolism and nutrition disorders) | 1 (2) | 2 (4) | 0 (0)
Elevated Amylase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated Creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated Lipase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 9 (13) | 2 (2) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hernia Repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 5 (6) | 0 (0) | 3 (3)
Left Ventricular Diastolic Dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pain (General disorders) | 2 (2) | 0 (0) | 2 (2)
Peripharal Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Prolonged QTc interval (Cardiac disorders) | 2 (3) | 0 (0) | 1 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Retinoic acid syndrome (Investigations) | 4 (4) | 2 (2) | 1 (1)
Sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATRA + ATO: Low Risk (WBC<10,000) (N=57) | ATRA+ATO+IDA: High Risk (WBC >10,000) (N=5) | ATO+ATRA+GO (N=16)
Infection (Infections and infestations) | 5 (5) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes